CLINICAL TRIAL: NCT04905004
Title: Comparing Canine Retraction Using Two-week, Four-week, Six-week and Eight-week Reactivation Intervals
Brief Title: Efficiency of Canine Retraction Using Different Reactivation Intervals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Yehya Mostafa, Head of the Orthodontics Department, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20153110-8-14-2017
Record Dates: First submitted 2021-05-23; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Class II Division 1 Malocclusion; Class III Malocclusion; Bimaxillary Protrusion; Crowding, Tooth
MeSH Terms: conditions — Malocclusion, Angle Class II; Malocclusion, Angle Class III; Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2-week reactivation interval (Experimental): Replacement of elastomeric chain every 2 weeks and reestablishing a 150 g force
  Interventions: Procedure: Canine retraction
- 4-week reactivation interval (Active Comparator): Replacement of elastomeric chain every 4 weeks and reestablishing a 150 g force
  Interventions: Procedure: Canine retraction
- 6-week reactivation interval (Experimental): Replacement of elastomeric chain every 6 weeks and reestablishing a 150 g force
  Interventions: Procedure: Canine retraction
- 8-week reactivation interval (Experimental): Replacement of elastomeric chain every 8 weeks and reestablishing a 150 g force
  Interventions: Procedure: Canine retraction

INTERVENTIONS:
Procedure: Canine retraction — Canines will be retracted using short elastomeric chains. Force applied to canines will be 150g.

SUMMARY:
Canine retraction after 1st premolar extracion into the extraction space is a routine treatment in orthodontics. Orthodontic patients requiring first premolar extraction, canine retraction and maximum anchorage were recruited for this randomized controlled trial. A search of the literature did not indicate the ideal frequency of elastomeric chain reactivation for optimum canine retraction. The study was approved by the ethical committee. The first premolars were extracted. Elastomeric chains were used to retract the canine distally into the 1st premolar space. The optimum reactivation interval was evaluated regarding the efficiency of treatment in terms of rate of canine retraction, canine tipping and rotation, root resorption and pain at the intervals of 2, 4, 6 and 8 weeks. Three dimensional imaging, as well as digital scanning were the methods for data collection.

DETAILED DESCRIPTION:
The canines, 2nd premolars, 1st molars and 2nd molars were bonded and banded. Leveling and alignment was achieved. After the first premolar extraction, temporary anchorage devices were inserted interradicular between 2nd premolar and 1st molar. Canine retraction was performed on a 0.016" X 0.022" stainless steel arch wire. A power arm was extended to apply the force closer to the center of resistance and achieve bodily movement. Elastomeric chains were calibrated to deliver a force of 150g and extended from the power arm to the mini screws directly. Recruited patients were randomly allocated to four groups according to the duration between the elastomeric chain reactivation. Canine reactivation intervals were 2, 4, 6, or 8 weeks. Cone beam computed tomography was performed before canine retraction and after 6 months of retraction. Digital dental casts were taken before canine retraction and monthly for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring 1st premolar extraction (e.g bimaxillary dentoalveolar protrusion)
* Erupted full set of permanent teeth (excluding 3rd molars)

Exclusion Criteria:

* Systemic diseases that would interfere with bone metabolism
* Craniofacial syndromes
* congenitally missing or extracted permanent teeth.
* periodontally compromised patients
* smokers
* pregnant women
* previous orthodontic treatment

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of canine retraction | Baseline to 1 month
  The distance measured between the canine cusp tips for each two consecutive digital models superimposed on the right and left medial palatal rugae.
Rate of canine retraction | 1month to 2 months
  The distance measured between the canine cusp tips for each two consecutive digital models superimposed on the right and left medial palatal rugae.
Rate of canine retraction | 2 months to 3 months
  The distance measured between the canine cusp tips for each two consecutive digital models superimposed on the right and left medial palatal rugae.
Rate of canine retraction | 3 months to 4 months
  The distance measured between the canine cusp tips for each two consecutive digital models superimposed on the right and left medial palatal rugae.
Rate of canine retraction | 4 months to 5 months
  The distance measured between the canine cusp tips for each two consecutive digital models superimposed on the right and left medial palatal rugae.
Rate of canine retraction | 5 months to 6 months.
  The distance measured between the canine cusp tips for each two consecutive digital models superimposed on the right and left medial palatal rugae.

SECONDARY OUTCOMES:
Amount of canine retraction | Baseline to 6 months
  The change in distance measured from the canine cusp tip to the frontal plane, in millimeters; measured on CBCT
Canine tipping | Baseline to 6 months
  CBCT images at T0 and T1 were analyzed using Invivo 5 software. linear measurements were made from the long axis of the canines (cusp tip to root apex) to FP1 and FP2 for the upper and lower canines, respectively.
Canine rotation | Baseline to 6 months
  The change in the angle between a line connecting the maximum mesial and distal crown convexities and FP1 and FP2, for the upper and lower canines, respectively; measured on CBCT
Canine root resorption | Baseline to 6 months
  The change in the canine length, in millimeters, measured from cusp tip to root apex; measured on CBCT
First molar anchorage loss | Baseline to 6 months
  The change in distance measured from the mesio-buccal cusp tip of the first molar to the frontal plane, in millimeters; measured on CBCT
Pain score | baseline to day 1
  The patient makes a mark along the Visual Analogue Scale (VAS) scale denoting the severity of pain: 0-100 0= no pain and 100= worst pain imaginable
Pain score | Baseline to day 2
  The patient makes a mark along the Visual Analogue Scale (VAS) scale denoting the severity of pain: 0-100 0= no pain and 100= worst pain imaginable
Pain score | Baseline to day 3
  The patient makes a mark along the Visual Analogue Scale (VAS) scale denoting the severity of pain: 0-100 0= no pain and 100= worst pain imaginable
Pain score | Baseline to day 4
  The patient makes a mark along the Visual Analogue Scale (VAS) scale denoting the severity of pain: 0-100 0= no pain and 100= worst pain imaginable
Pain score | Baseline to day 5
  The patient makes a mark along the Visual Analogue Scale (VAS) scale denoting the severity of pain: 0-100 0= no pain and 100= worst pain imaginable
Pain score | Baseline to day 6
  The patient makes a mark along the Visual Analogue Scale (VAS) scale denoting the severity of pain: 0-100 0= no pain and 100= worst pain imaginable
Pain score | Baseline to day 7
  The patient makes a mark along the Visual Analogue Scale (VAS) scale denoting the severity of pain: 0-100 0= no pain and 100= worst pain imaginable
Pain score | Baseline to day 8
  The patient makes a mark along the Visual Analogue Scale (VAS) scale denoting the severity of pain: 0-100 0= no pain and 100= worst pain imaginable
Pain score | Baseline to day 9
  The patient makes a mark along the Visual Analogue Scale (VAS) scale denoting the severity of pain: 0-100 0= no pain and 100= worst pain imaginable
Pain score | Baseline to day 10.
  The patient makes a mark along the Visual Analogue Scale (VAS) scale denoting the severity of pain: 0-100 0= no pain and 100= worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Yehya Mostafa, PhD, Study Director — Future University in Egypt
Locations (1):
- Future University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No